CLINICAL TRIAL: NCT02321436
Title: Asian Multicentre, Double Blind, Randomised, Placebo Controlled Pilot Study, to Assess the Impact of Dysport® Intramuscular Injections When Administered Within the First 12 Weeks After Stroke on the Time to Spasticity Progression in Adult Subjects With Upper Limb (UL) Spasticity.
Brief Title: Study to Assess Impact of Dysport Injections Early After Stroke on Upper Limb Spasticity Progression
Acronym: ONTIME Pilot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-79-52120-197
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Upper Limb Spasticity
MeSH Terms: conditions — Stroke | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Active Comparator): Dysport® 500U intramuscular injection
  Interventions: Biological: Botulinum toxin type A
- Placebo Group (Placebo Comparator): Placebo intramuscular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Botulinum toxin type A — Subjects to receive Dysport® 500U administered intramuscularly in the targeted upper limb.
  Other Names: AbobotulinumtoxinA (Dysport®)
  Arms: Treatment group
Drug: Placebo — Placebo administered intramuscularly in the targeted upper limb.
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to investigate if early administration (i.e. within 12 weeks after stroke) of Dysport® 500 U injections may delay the appearance or the progression of upper limb symptomatic spasticity.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 12 weeks after first ever stroke according to the World Health Organisation criteria (previous transient ischaemic attack or clinically silent infarct on computerised tomography (CT)/magnetic resonance imaging (MRI) are not counted as previous stroke)
* Stroke confirmed by CT/MRI scan and classified as ischaemic/haemorrhagic stroke
* Presence of spasticity:

  * either symptomatic, based on symptomatic spasticity criteria (i.e. at least one of the following items: impacted passive/active function, involuntary movements, or pain ≥4 on a numeric pain rating scale [NPRS]), in addition to increased muscle tone [Modified Ashworth Scale, MAS ≥2])
  * or only increased muscle tone (MAS≥2)

Exclusion Criteria:

* Neuromuscular junction (NMJ) diseases, or any other neurological disorders (including prior local joint, tendon, and intrinsic muscle disorders) that could potentially interfere with assessment of spasticity in the primary targeted muscle group selected by the Investigator and in agreement with the subject
* Currently receiving drugs affecting NMJ transmission e.g. aminoglycosides, aminoquinolines, cyclosporine, D penicillamine
* Previous surgery of the affected muscles/ ligaments/tendons
* Severe comorbidities (e.g. congestive heart failure, myocardial infarction, multiple organ failure, hepatic renal failures, severe infections)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (4):
- Neurology Laboratory -University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Center for Neurodiagnostic and Therapeutic Services Metropolitan Medical Center, Manila, Philippines
- TTSH Rehabilitation Centre Ang Mo Kio Community Hospital, Singapore, Singapore
- Department of rehabilitation Medicine Faculty of medicine Siriraj Hospital, Madihol University Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Rosales RL, Balcaitiene J, Berard H, Maisonobe P, Goh KJ, Kumthornthip W, Mazlan M, Latif LA, Delos Santos MMD, Chotiyarnwong C, Tanvijit P, Nuez O, Kong KH. Early AbobotulinumtoxinA (Dysport(R)) in Post-Stroke Adult Upper Limb Spasticity: ONTIME Pilot Study. Toxins (Basel). 2018 Jun 21;10(7):253. doi: 10.3390/toxins10070253. PMID 29933562

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 adult subjects with upper limb (UL) spasticity were enrolled into a multicentre, prospective, double-bind, randomised, placebo-controlled pilot study, conducted in four countries (Malaysia, Thailand, Singapore, and the Philippines).
Pre-assignment Details: The first visit was scheduled within 2 to 12 weeks post-stroke and subjects were randomized at a ratio of 2:1 to receive either Dysport® 500 Units (U) or placebo. Dysport® was expected to have a beneficial effect in these subjects so the unbalanced randomisation ratio was chosen in order to expose the minimum number of subjects to inactive placebo.
Groups:
- Dysport ® 500 U: Dysport® 500 U was administered at the clinic in a single intramuscular (IM) injection in the targeted UL. The investigator was allowed to adjust the dose per targeted muscle, depending on the level of hypertonicity, as long as the total fixed dosage per subject was 500 U/2.5 millilitre (mL).
  Evaluation of reinjection criteria started at Week 4 post-injection of Dysport®. Assessments were then performed every 2 weeks until Week 12. Following Week 12, assessments were performed every 4 weeks until Week 28. The subject's last study visit was the visit when reinjection criteria was met, Week 28, or early withdrawal visit.
- Placebo: Placebo was administered at the clinic in a single IM injection in the targeted UL. Evaluation of reinjection criteria started at Week 4 post-injection of placebo. Assessments were then performed every 2 weeks until Week 12. Following Week 12, assessments were performed every 4 weeks until Week 28. The subject's last study visit was the visit when reinjection criteria was met, Week 28, or early withdrawal visit.
Period: Overall Study
Arm/Group | Dysport ® 500 U | Placebo
Started | 28 | 14
Completed | 27 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the 42 subjects with UL spasticity who were enrolled and treated with either Dysport® 500 U or placebo.
Groups:
- Dysport ® 500 U: Dysport® 500 U was administered at the clinic in a single IM injection in the targeted UL. The investigator was allowed to adjust the dose per targeted muscle, depending on the level of hypertonicity, as long as the total fixed dosage per subject was 500 U/2.5 mL.
  Evaluation of reinjection criteria started at Week 4 post-injection of Dysport®. Assessments were then performed every 2 weeks until Week 12, Following Week 12, assessments were performed every 4 weeks until Week 28. The subject's last study visit was the visit when reinjection criteria was met, Week 28, or early withdrawal visit.
Arm/Group | Dysport ® 500 U | Placebo | Total Title
Number analyzed (Participants) | 28 | 14 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (13.2) | 56.5 (9.7) | 59.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 23 | 10 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 28 | 14 | 42
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Country [Number; unit: Participants]
  Malaysia | 3 | 1 | 4
  Philippines | 11 | 4 | 15
  Singapore | 9 | 5 | 14
  Thailand | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Time Between the Initial Injection and the Appearance of Reinjection Criteria as Evaluated by the Modified Ashworth Scale (MAS) and Spasticity Symptoms
Description: The appearance of increased muscle tone was assessed using the MAS (scale ranges from 0 [no increase in muscle tone] to 4 [affected part rigid in flexion or extension]). For confirmation of reinjection criteria appearance, a subject had to have a MAS score in the primary targeted muscle group of ≥2 and at least 1 of the following 4 criteria confirming signs of symptomatic spasticity in the UL:
  1. A Numeric Pain Rating Scale (NPRS) pain score ≥ 4 (NPRS ranges from 0 [no pain] to 10 [severe pain])
  2. An impact on passive function measured by a score of ≥ 1 on the 4-point Likert scale (scale ranges from 0 [no impact] to 3 [severe impact])
  3. An impact on active function measured by a score of ≥ 1 on the 4-point Likert scale
  4. An involuntary movements score ≥1 on the 4-point Likert scale in relevant upper limb.
  Results are reported overall for subjects with both symptomatic and asymptomatic spasticity.
Time Frame: From Week 4 up to Week 28
Population: This analysis was performed on the Intention-To-Treat (ITT) population which includes all randomised subjects who provided informed consent.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dysport ® 500 U | Placebo
Number analyzed (Participants) | 28 | 14
days | 156 [86 to 206] | 32 [29 to 114]
Statistical Analysis 1: Comparison: Dysport ® 500 U vs Placebo; Test type: Other — The treatment difference (Dysport® versus placebo) was tested using a non-parametric, two-sided, stratified log rank test; p = 0.0176, Log Rank — Significance level (α) = 5%
Statistical Analysis 2: Comparison: Dysport ® 500 U vs Placebo; Test type: Other — The treatment difference (Dysport® versus placebo) was tested using a non-parametric, two-sided, stratified Wilcoxon test; p = 0.0480, Wilcoxon (Mann-Whitney) — Significance level (α) = 5%

2. Secondary Outcome: Mean Change in MAS of the Primary Targeted Muscle Group.
Description: Increased muscle tone in the primary muscle group (selected by the investigator at the first visit, based on his/her clinical judgement and in agreement with the subject, in one of the following muscle groups: elbow flexors or pronators, wrist flexors, or finger flexors) was assessed using the MAS. Scale ranges from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension). Least Squares (LS) mean change from baseline to each subsequent visit (including the subject's last study visit) of the MAS score is reported.
Time Frame: From baseline up to Week 28
Population: This analysis was performed on the ITT population which includes all randomised subjects who provided informed consent.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Dysport ® 500 U | Placebo
Number analyzed (Participants) | 28 | 14
units on a scale
  Visit 2 (Week 4) | -1.27 (0.17) | -0.26 (0.22)
  Visit 3 (Week 6) | -1.29 (0.19) | -0.24 (0.24)
  Visit 4 (Week 8): number analyzed (Participants) | 27 | 13
  Visit 4 (Week 8) | -1.29 (0.18) | -0.24 (0.24)
  Visit 5 (Week 10): number analyzed (Participants) | 28 | 13
  Visit 5 (Week 10) | -1.06 (0.17) | -0.22 (0.22)
  Visit 6 (Week12): number analyzed (Participants) | 28 | 13
  Visit 6 (Week12) | -0.86 (0.18) | -0.03 (0.24)
  Visit 7 (Week 16): number analyzed (Participants) | 18 | 4
  Visit 7 (Week 16) | -1.14 (0.18) | -0.63 (0.35)
  Visit 8 (Week 20): number analyzed (Participants) | 14 | 2
  Visit 8 (Week 20) | -0.9 (0.19) | -0.75 (0.47)
  Visit 9 (Week 24): number analyzed (Participants) | 13 | 2
  Visit 9 (Week 24) | -0.87 (0.24) | -0.75 (0.57)
  Visit 10 (Week 28): number analyzed (Participants) | 12 | 2
  Visit 10 (Week 28) | -0.96 (0.2) | -0.75 (0.42)
Statistical Analysis 1: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 2 (Week 4); Test type: Other — Differences between treatment groups and p-values are based on an analysis of variance performed at each visit, taking into account treatment and spasticity status as fixed effects. Baseline value is value assessed at Visit 1; p = 0.0005, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -1.00, 95% CI 2-sided [-1.54 to -0.47]
Statistical Analysis 2: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 3 (Week 6); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0007, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.63 to -0.47]
Statistical Analysis 3: Comparison: Dysport ® 500 U; Differences between treatment groups at Visit 4 (Week 8); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0006, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -1.05, 95% CI 2-sided [-1.62 to -0.48]
Statistical Analysis 4: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 5 (Week 10); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0027, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.36 to -0.31]
Statistical Analysis 5: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 6 (Week 12); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0052, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.39 to -0.26]
Statistical Analysis 6: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 7 (Week 16); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2037, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-1.35 to 0.31]
Statistical Analysis 7: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 8 (Week 20); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.7656, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-1.25 to 0.94]
Statistical Analysis 8: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 9 (Week 24); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.8521, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-1.46 to 1.23]
Statistical Analysis 9: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 10 (Week 28); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.6582, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.24 to 0.81]

3. Secondary Outcome: Mean Change in Fugl-Meyer Assessment for Evaluation of UL Motor Impairment.
Description: The Fugl-Meyer assessment is a validated tool for measuring motor functioning, balance, sensation, and joint functioning in the upper or lower limbs of subjects with post-stroke hemiplegia. The assessment scale is comprised of 155 items across 5 domains: motor functioning, sensory functioning, balance, joint range of motion and joint pain. For this study, only the UL motor part was assessed using the following criteria:
  A. Upper Extremity (from 0 to 36) B. Wrist (from 0 to 10) C. Hand (from 0 to 14) D. Coordination / Speed (from 0 to 6)
  Total motor function scores (A-D [from 0 to 66]) were calculated and LS mean changes from baseline up to (but not including) the visit when the reinjection criteria were met were reported.
  Higher values for change from baseline indicated a better outcome.
Time Frame: From baseline up to Week 28
Population: This analysis was performed on the ITT population and includes all randomised subjects who provided informed consent.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Dysport ® 500 U: Dysport® 500 U was administered at the clinic in a single IM injection in the targeted UL. The investigator was allowed to adjust the dose per targeted muscle, depending on the level of hypertonicity, as long as the total fixed dosage per subject was 500 U/2.5mL.
  Evaluation of reinjection criteria started at Week 4 post-injection of Dysport®. Assessments were then performed every 2 weeks until Week 12, Following Week 12, assessments were performed every 4 weeks until Week 28. The subject's last study visit was the visit when reinjection criteria was met, Week 28, or early withdrawal visit.
Arm/Group | Dysport ® 500 U | Placebo
Number analyzed (Participants) | 28 | 14
units on a scale
  Visit 2 (Week 4): number analyzed (Participants) | 22 | 6
  Visit 2 (Week 4) | 6.4 (2.5) | 5.6 (4.4)
  Visit 3 (Week 6): number analyzed (Participants) | 22 | 5
  Visit 3 (Week 6) | 7.4 (2.6) | 8.3 (5.0)
  Visit 4 (Week 8): number analyzed (Participants) | 22 | 5
  Visit 4 (Week 8) | 6.9 (2.6) | 9.2 (5.0)
  Visit 5 (Week 10): number analyzed (Participants) | 21 | 5
  Visit 5 (Week 10) | 10.3 (2.9) | 10.4 (5.4)
  Visit 6 (Week 12): number analyzed (Participants) | 18 | 4
  Visit 6 (Week 12) | 11.1 (3.5) | 6.5 (6.9)
  Visit 7 (Week 16): number analyzed (Participants) | 15 | 2
  Visit 7 (Week 16) | 9.4 (3.7) | 21.8 (9.2)
  Visit 8 (Week 20): number analyzed (Participants) | 14 | 2
  Visit 8 (Week 20) | 9.4 (4.4) | 23.5 (10.5)
  Visit 9 (Week 24): number analyzed (Participants) | 12 | 2
  Visit 9 (Week 24) | 14.8 (4.6) | 23.8 (9.8)
  Visit 10 (Week 28): number analyzed (Participants) | 11 | 2
  Visit 10 (Week 28) | 15.0 (5.4) | 19.5 (11.5)
Statistical Analysis 1: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 2 (Week 4); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.8754, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-9.5 to 11.1]
Statistical Analysis 2: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 3 (Week 6); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.8805, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-12.8 to 11.1]
Statistical Analysis 3: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 4 (Week 8); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.6992, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-14.0 to 9.6]
Statistical Analysis 4: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 5 (Week 10); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.9882, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-13.0 to 12.8]
Statistical Analysis 5: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 6 (Week 12); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.5646, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-11.9 to 21.2]
Statistical Analysis 6: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 7 (Week 16); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2325, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -12.5, 95% CI 2-sided [-34.0 to 9.0]
Statistical Analysis 7: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 8 (Week 20); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2441, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -14.1, 95% CI 2-sided [-39.4 to 11.1]
Statistical Analysis 8: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 9 (Week 24); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.4311, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -9.0, 95% CI 2-sided [-33.7 to 15.7]
Statistical Analysis 9: Comparison: Dysport ® 500 U vs Placebo; Differences between treatment groups at Visit 10 (Week 28); Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.7310, ANOVA — p value significance level = 5%; Mean Difference (Final Values) = -4.5, 95% CI 2-sided [-33.3 to 24.3]

4. Secondary Outcome: Global Assessment of Changes at Last Visit
Description: Global assessment of changes was assessed by the investigator from Week 4 up to (but not including) the visit when the reinjection criteria were met. This endpoint was assessed by the investigator using a 5-point Likert scale to answer the following question: How does your patient feel compared to his/her condition at the first visit?
  * Much better
  * Better
  * No change
  * Worse
  * Much worse
  Results are reported overall for subjects with both symptomatic and asymptomatic spasticity.
Time Frame: From Week 4 up to Week 28
Population: This efficacy analysis was performed on the ITT population which includes all randomised subjects who provided informed consent. No data is available for subjects who met their reinjection criteria at Visit 2 (Week 4).
Measure: Number; unit: percentage of participants
Arm/Group | Dysport ® 500 U | Placebo
Number analyzed (Participants) | 22 | 6
percentage of participants
  Much Better | 9.1 | 0
  Better | 81.8 | 83.3
  No Change | 4.5 | 16.7
  Worse | 4.5 | 0
  Much Worse | 0 | 0
Statistical Analysis 1: Comparison: Dysport ® 500 U vs Placebo; Test type: Other; p = 0.6128, Cochran-Mantel-Haenszel — The Cochran-Mantel-Haenszel (CMH) p-value represents the strength of the association between treatment and global assessments of changes at the last visit, adjusted for symptomatic status at baseline; p value significance level = 5%

5. Secondary Outcome: Number of Concomitant Non-drug Therapy Sessions.
Description: The number of non-drug therapy sessions that the subject received for UL spasticity in combination with injections of either Dysport® or placebo - up to and including the subject's last study visit - were recorded in the Electronic Case Report Form (eCRF) as part of concomitant medications and therapies evaluation at all study visits (Prior and Concomitant Non-Drug Therapies eCRF page). All concomitant therapies in the indication of "Post Stroke UL Spasticity" were counted by subject from first administration of Dysport® or placebo to last study visit. Concomitant non-drug therapies were defined as received any time during study (on or after the day of the first injection of Dysport® or placebo) regardless of the start or stop date. For each subject, overlapping sessions were defined as one therapy session using the earliest start date as the start date and the latest start date as the stop date.
Time Frame: From baseline up to Week 28
Population: This analysis was performed on the safety population which includes all randomised subjects who received the study medication.
Measure: Number; unit: Number of sessions
Arm/Group | Dysport ® 500 U | Placebo
Number analyzed (Participants) | 28 | 14
Number of sessions
  Any concomitant non-drug therapies | 25 | 14
  Physiotherapy | 22 | 14
  Other therapies | 8 | 5

6. Secondary Outcome: Mean Duration of Concomitant Non-drug Therapy Sessions.
Description: The duration of non-drug therapy sessions that the subject received for UL spasticity in combination with injections of either Dysport® or placebo - up to and including the subject's last study visit - were recorded in the Electronic Case Report Form (eCRF) as part of concomitant medications and therapies evaluation at all study visits (Prior and Concomitant Non-Drug Therapies eCRF page). Overall duration of concomitant therapies in the indication of "Post Stroke UL Spasticity" was computed for the period from first administration of Dysport® or placebo to last study visit. Concomitant non-drug therapies were defined as received any time during study (on or after the day of the first injection of Dysport® or placebo) regardless of the start or stop date. For each subject, overlapping sessions were defined as one therapy session using the earliest start date as the start date and the latest start date as the stop date.
Time Frame: From baseline up to Week 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dysport ® 500 U | Placebo
Number analyzed (Participants) | 28 | 14
days
  Any concomitant non-drug therapies | 160.5 (56.8) | 126.1 (55.0)
  Physiotherapy | 157.9 (59.2) | 126.1 (55.0)
  Other therapies | 184.9 (41.3) | 154.6 (84.4)

ADVERSE EVENTS:
Time Frame: Up to Week 28.
Description: Treatment Emergent Adverse Events (TEAEs) were reported and defined as any Adverse Event (AE) that emerged or worsened during the active phase of the study.
Arm/Group | Dysport ® 500 U | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/14
Serious Adverse Events (participants affected / at risk) | 3/28 | 0/14
Other Adverse Events (participants affected / at risk) | 5/28 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport ® 500 U (N=28) | Placebo (N=14)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dysport ® 500 U (N=28) | Placebo (N=14)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the first communication or publication regarding the study must be a joint publication between the PI and Sponsor.